CLINICAL TRIAL: NCT02357459
Title: A Double-Blind, Randomized, Single-Dose Study to Assess the Safety and Efficacy of FX006 for the Treatment of Pain in Patients With Osteoarthritis of the Knee
Brief Title: Study of FX006 for the Treatment of Pain in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2014-008
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; pain; corticosteroid; intra-articular; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006; Triamcinolone; Saline Solution; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FX006 32mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release Formulation
  Interventions: Drug: FX006
- Normal Saline (Placebo Comparator): Single 5 mL intra-articular (IA) injection
  Interventions: Drug: Placebo
- TCA IR 40 mg (Active Comparator): Single 1 mL intra-articular (IA) injection TCA IR 40 mg: Immediate-release formulation
  Interventions: Drug: TCA IR 40

INTERVENTIONS:
Drug: FX006 — Single 5 mL IA injection
  Other Names: Zilretta
  Arms: FX006 32mg
Drug: Placebo — Single 5 mL IA injection
  Other Names: Normal Saline
  Arms: Normal Saline
Drug: TCA IR 40 — Single 1 mL IA injection
  Other Names: Kenalog®-40 Injection; Kenacort-A 40; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
The purpose of this study was to assess the safety and efficacy of FX006 for the treatment of pain in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This study was a double-blind, randomized, single dose design. The study was conducted in male and female patients ≥40 years of age with OA of the knee. Approximately 450 patients with OA of the knee were randomized to 1 of 3 treatment groups (1:1:1) and treated with a single IA injection of:

* 32 mg FX006,
* normal saline (placebo), or
* 40 mg TCA IR.

Randomization was stratified by weekly mean of the average daily (24-hour) pain intensity (ADP) scores at baseline, with the following classifications: 5 to <6, 6 to <7, and ≥7.

Each patient was evaluated for a total of 24 weeks following a single IA injection. Following screening, safety and efficacy were evaluated at 7 out-patient visits (Days 1 [baseline], Weeks 4, 8, 12, 16, 20, and 24). The study was expected to enroll in approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female >=40 years of age
* Has symptoms associated with OA of the index knee for at least 6 months prior to Screening
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA
* Kellgren-Lawrence (K-L) Grade 2 or 3 in the index knee per Screening X-ray
* Index knee pain for > 15 days over the last month
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of restricted medications

Exclusion Criteria:

* Any condition that could possibly confound the patient's assessment of index knee pain in judgement of the investigator (i.e., iIpsilateral hip OA, gout, radicular low back pain and hip pain that is referred to the knee that could cause misclassification, pain in any other area of the lower extremities or back that is equal or greater than the index knee pain)
* Fibromyalgia, Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease
* History of infection in the index knee
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee within 1 month of Screening
* Unstable joint within 12 months of screening
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Intramuscular (IM) or oral corticosteroids (investigational or marketed) within 1 month of Screening
* Any other IA investigational drug/biologic within 6 months of Screening
* Prior use of FX006
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (37):
- United States (21):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Canoga Park, California
  - North Hollywood, California
  - San Diego, California
  - Denver, Colorado
  - Atlantis, Florida
  - DeLand, Florida
  - Hialeah, Florida
  - Sarasota, Florida
  - West Palm Beach, Florida
  - Prairie Village, Kansas
  - Albuquerque, New Mexico
  - Cary, North Carolina
  - PMG Research of Cary, Cary, North Carolina
  - Charlotte, North Carolina
  - Duncansville, Pennsylvania
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Dallas, Texas
  - Newport News, Virginia
- Australia (6):
  - Broadmeadow, New South Wales
  - Geelong, New South Wales
  - Merewether, New South Wales
  - St Leonards, New South Wales
  - Sherwood, Queensland
  - Malvern, Victoria
- Canada (3):
  - Quebec, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Tallinn, Estonia
- Hong Kong, Hong Kong
- Vilnius, Lithuania
- Bucharest, Romania

REFERENCES:
- [Derived] Ross E, Katz NP, Conaghan PG, Kivitz A, Turk DC, Spitzer AI, Jones DG, Lanier RK, Cinar A, Lufkin J, Kelley SD. Improved Treatment Effect of Triamcinolone Acetonide Extended-Release in Patients with Concordant Baseline Pain Scores on the Average Daily Pain and Western Ontario and McMaster Universities Osteoarthritis Index Pain Scales. Pain Ther. 2022 Mar;11(1):289-302. doi: 10.1007/s40122-021-00335-z. Epub 2021 Nov 17. PMID 34791634
- [Derived] Langworthy MJ, Conaghan PG, Ruane JJ, Kivitz AJ, Lufkin J, Cinar A, Kelley SD. Efficacy of Triamcinolone Acetonide Extended-Release in Participants with Unilateral Knee Osteoarthritis: A Post Hoc Analysis. Adv Ther. 2019 Jun;36(6):1398-1411. doi: 10.1007/s12325-019-00944-3. Epub 2019 Apr 9. PMID 30968336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at 41 centers across the United States, Canada, Australia, New Zealand, Hong Kong, Denmark, Romania, Estonia and Lithuania. Enrollment took approximately 6 months
Pre-assignment Details: Subjects were screened within 21 days of being randomized.
Groups:
- FX006 32mg: 161 subjects received FX006 32 mg as a single 5 mL IA injection
- Placebo: 162 subjects received normal saline as a single 5 mL IA injection.
- TCA IR 40 mg: 161 subjects received TCA IR 40 mg as a single 1 mL IA injection
Period: Overall Study
Arm/Group | FX006 32mg | Placebo | TCA IR 40 mg
Started | 161 | 163 | 162
Completed | 144 | 149 | 150
Not Completed | 17 | 14 | 12
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 3
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Lack of Efficacy | 7 | 4 | 4
Not completed — Patient Relocated | 2 | 0 | 0
Not completed — Instruction from PCP | 1 | 0 | 0
Not completed — Incarceration | 0 | 0 | 1
Not completed — Pre-planned Knee surgery | 0 | 0 | 2
Not completed — Job Commitments | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 486 patients were randomized in the study. Two patients, 1 each in the placebo group and 40 mg TCA IR group, were randomized and not treated. These 2 patients were not included in the FAS, Safety, or PP populations.
Groups:
- Placebo: Normal Saline: Single 5 mL IA injection
- TCA IR 40 mg: TCA IR: Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 32mg | Placebo | TCA IR 40 mg | Total
Number analyzed (Participants) | 161 | 162 | 161 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.52) | 62.4 (8.89) | 62.3 (10.08) | 62.1 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 96 | 97 | 296
  Male | 58 | 66 | 64 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Mean of the Average Daily (24-hr) Pain (ADP) Intensity Scores for 32 mg FX006 Versus Placebo
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where ) indicates "no pain" and 10 indicates "pain as bad as you can imagine."
Time Frame: Baseline and 12 Weeks
Population: Randomized patients who received study drug assigned to the FX006 32 mg arm and the placebo arm.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32mg | Placebo
Number analyzed (Participants) | 161 | 162
units on a scale | -3.12 (0.203) | -2.14 (0.202)
Statistical Analysis 1: Comparison: FX006 32mg vs Placebo; Test type: Superiority — The analysis included all study weeks of data, and was not confined to only that at Baseline and Week 12. Descriptive statistics included number of observations, unadjusted mean, standard deviation, median, minimum and maximum, and baseline adjusted means from the mixed model. Treatment differences from control was presented, and estimated via least squares means from the analysis model along with 95% confidence intervals and associated 2-sided p-values; p < 0.0001, longitudinal mixed repeated measures — The threshold for significance was <0.05; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.47 to -0.49], Standard Error of Mean 0.20

2. Secondary Outcome: Area Under the Effect Curve (AUE) of Change From Baseline in the Weekly Mean of the ADP Scores From Baseline to Week 12 for FX006 Relative to Placebo
Description: as for outcome 1
Time Frame: Baseline to 12 Weeks
Population: Randomized patients who received study drug assigned to the FX006 32 mg arm and the placebo arm
Measure: Least Squares Mean (Standard Error); unit: ADP Pain Scores * Week
Arm/Group | FX006 32mg | Placebo
Number analyzed (Participants) | 161 | 162
ADP Pain Scores * Week | -247.3 (14.89) | -145.3 (14.77)

3. Secondary Outcome: AUE of Change From Baseline in Weekly Mean of the ADP Scores From Baseline to Week 12 for FX006 Relative to TCA IR
Description: as for outcome 1
Time Frame: Baseline to 12 Weeks
Measure: Least Squares Mean (Standard Error); unit: ADP Pain Scores * Week
Groups:
- FX006 32 mg: FX006: Single 5 mL IA injection
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 161 | 161
ADP Pain Scores * Week | -247.3 (14.89) | -231.9 (14.85)

4. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Mean of the ADP Scores From Baseline to Week 12 for FX006 Relative to TCA IR
Description: as for outcome 1
Time Frame: Baseline through 12 Weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 161 | 161
units on a scale | -3.12 (0.203) | -2.86 (0.202)

5. Secondary Outcome: AUE of Change From Baseline in Weekly Mean of the ADP Scores From Baseline to Week 24 for FX006 Relative to Placebo
Description: as for outcome 1
Time Frame: Baseline to 24 Weeks
Population: AUE of Change From Baseline in Weekly Mean of the ADP Scores From Baseline to Week 24 for TCA IR 40 mg Relative to Placebo was not a pre-specified Secondary Outcome and therefore not reported
Measure: Least Squares Mean (Standard Error); unit: ADP Pain Scores * Week
Arm/Group | FX006 32mg | Placebo
Number analyzed (Participants) | 161 | 162
ADP Pain Scores * Week | -432.5 (30.14) | -297.0 (29.90)

6. Other Pre Specified Outcome: Change From Baseline to Each Week in Weekly Mean of the ADP Scores
Description: as for outcome 1
Time Frame: Weeks 1-11 & Weeks 13-24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
units on a scale
  Week 1 | -1.9 (0.202) | -1.04 (0.200) | -2.13 (0.201)
  Week 2 | -2.95 (0.202) | -1.61 (0.201) | -2.69 (0.201)
  Week 3 | -3.20 (0.202) | -1.66 (0.201) | -2.93 (0.202)
  Week 4 | -3.23 (0.202) | -1.84 (0.200) | -3.11 (0.202)
  Week 5 | -3.34 (0.202) | -1.87 (0.201) | -3.11 (0.202)
  Week 6 | -3.48 (0.202) | -1.95 (0.201) | -3.20 (0.202)
  Week 7 | -3.48 (0.202) | -2.01 (0.201) | -3.03 (0.202)
  Week 8 | -3.48 (0.202) | -1.96 (0.202) | -3.04 (0.202)
  Week 9 | -3.45 (0.202) | -2.06 (0.202) | -3.06 (0.202)
  Week 10 | -3.31 (0.202) | -2.08 (0.201) | -3.07 (0.202)
  Week 11 | -3.21 (0.203) | -2.13 (0.202) | -3.01 (0.202)
  Week 13 | -2.96 (0.203) | -2.21 (0.202) | -2.87 (0.202)
  Week 14 | -2.91 (0.203) | -2.18 (0.202) | -2.73 (0.202)
  Week 15 | -2.84 (0.204) | -2.12 (0.202) | -2.75 (0.202)
  Week 16 | -2.73 (0.204) | -2.22 (0.203) | -2.67 (0.203)
  Week 17 | -2.66 (0.204) | -2.18 (0.203) | -2.57 (0.203)
  Week 18 | -2.60 (0.204) | -2.13 (0.203) | -2.55 (.0203)
  Week 19 | -2.57 (0.204) | -2.19 (0.203) | -2.48 (0.202)
  Week 20 | -2.44 (0.204) | -2.18 (0.203) | -2.46 (0.202)
  Week 21 | -2.27 (0.204) | -2.16 (0.203) | -2.27 (0.203)
  Week 22 | -2.18 (0.205) | -2.20 (0.204) | -2.29 (0.203)
  Week 23 | -2.14 (0.205) | -2.12 (0.204) | -2.30 (0.203)
  Week 24 | -1.99 (0.205) | -2.16 (0.203) | -2.18 (0.203)

7. Other Pre Specified Outcome: Change From Baseline Over Time for WOMAC A (Pain Subscale) at Weeks 4, 8, 12, 16, 20 and 24.
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
units on a scale
  Week 4 | -1.10 (0.068) | -0.50 (0.067) | -0.87 (0.067)
  Week 8 | -1.02 (0.071) | -0.48 (0.070) | -0.81 (0.070)
  Week 12 | -0.88 (0.071) | -0.50 (0.071) | -0.70 (0.070)
  Week 16 | -0.67 (0.072) | -0.54 (0.071) | -0.64 (0.071)
  Week 20 | -0.61 (0.069) | -0.51 (0.069) | -0.60 (0.068)
  Week 24 | -0.63 (0.070) | -0.49 (0.070) | -0.56 (0.069)

8. Other Pre Specified Outcome: Change From Baseline Over Time for WOMAC B (Stiffness Subscale) at Weeks 4, 8, 12, 16, 20 and 24
Description: as for outcome 7
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
units on a scale
  Week 4 | -1.23 (0.079) | -0.51 (0.077) | -1.00 (0.078)
  Week 8 | -1.24 (0.078) | -0.54 (0.077) | -0.92 (0.077)
  Week 12 | -1.03 (0.079) | -0.59 (0.078) | -0.80 (0.078)
  Week 16 | -0.80 (0.080) | -0.64 (0.080) | -0.71 (0.079)
  Week 20 | -0.66 (0.078) | -0.64 (0.078) | -0.58 (0.077)
  Week 24 | -0.67 (0.080) | -0.58 (0.079) | -0.57 (0.079)

9. Other Pre Specified Outcome: Change From Baseline Over Time for WOMAC C (Function Subscale) at Weeks 4, 8, 12, 16, 20 and 24
Description: as for outcome 7
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
units on a scale
  Week 4 | -1.11 (.066) | -0.51 (.065) | -0.87 (.065)
  Week 8 | -1.09 (.068) | -0.53 (.068) | -0.80 (.068)
  Week 12 | -0.93 (.069) | -0.56 (.068) | -0.72 (.068)
  Week 16 | -0.69 (.069) | -0.59 (.069) | -0.62 (.069)
  Week 20 | -0.65 (.068) | -0.56 (.068) | -0.57 (.067)
  Week 24 | -0.59 (.069) | -0.51 (.069) | -0.54 (.068)

10. Other Pre Specified Outcome: Change From Baseline Over Time for Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) Subscale at Weeks 4, 8, 12 and 24
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) is a participant (patient)-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury and also consequences of primary osteoarthritis (OA). It holds 42 items in five separately scored subscales: KOOS Pain, KOOS Symptoms, Function in daily living (KOOS ADL), Function in Sport and Recreation (KOOS Sport/Rec), and knee-related Quality of Life (KOOS QOL).
  A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). Each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Higher scores indicate better quality of life.
Time Frame: Weeks 4, 8, 12, and 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 136 | 144 | 134
units on a scale
  Week 4 | 23.50 (1.896) | 8.93 (1.832) | 15.60 (1.882)
  Week 8 | 23.30 (1.907) | 10.70 (1.856) | 18.02 (1.891)
  Week 12 | 21.19 (1.907) | 12.22 (1.869) | 15.77 (1.895)
  Week 24 | 11.95 (1.923) | 10.25 (1.878) | 11.44 (1.906)

11. Other Pre Specified Outcome: Responder Status as Defined by Proportion of Patients Experiencing >30% Decrease in Pain From Baseline in Weekly Mean of the ADP Scores at Each Week (Weeks 1-24)
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine."
Time Frame: Weeks 1-24
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
Participants
  Week 1 | 66 | 42 | 81
  Week 2 | 99 | 63 | 96
  Week 3 | 109 | 61 | 101
  Week 4 | 107 | 64 | 108
  Week 5 | 106 | 69 | 109
  Week 6 | 113 | 73 | 111
  Week 7 | 112 | 75 | 112
  Week 8 | 109 | 74 | 107
  Week 9 | 107 | 79 | 109
  Week 10 | 107 | 78 | 109
  Week 11 | 107 | 78 | 105
  Week 12 | 103 | 80 | 104
  Week 13 | 97 | 81 | 106
  Week 14 | 95 | 80 | 100
  Week 15 | 88 | 79 | 97
  Week 16 | 91 | 81 | 97
  Week 17 | 84 | 82 | 86
  Week 18 | 81 | 75 | 93
  Week 19 | 86 | 78 | 88
  Week 20 | 84 | 79 | 87
  Week 21 | 82 | 76 | 83
  Week 22 | 79 | 74 | 78
  Week 23 | 77 | 79 | 84
  Week 24 | 70 | 74 | 74

12. Other Pre Specified Outcome: Responder Status as Defined by Proportion of Patients Experiencing >50% Decrease in Pain From Baseline in Weekly Mean of the ADP Scores at Each Week (Weeks 1-24)
Time Frame: Weeks 1-24
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
Participants
  Week 1 | 39 | 21 | 57
  Week 2 | 73 | 37 | 67
  Week 3 | 81 | 40 | 77
  Week 4 | 86 | 47 | 80
  Week 5 | 85 | 51 | 80
  Week 6 | 92 | 51 | 84
  Week 7 | 97 | 49 | 85
  Week 8 | 97 | 53 | 82
  Week 9 | 91 | 55 | 83
  Week 10 | 87 | 57 | 84
  Week 11 | 83 | 60 | 80
  Week 12 | 80 | 56 | 75
  Week 13 | 79 | 57 | 77
  Week 14 | 76 | 54 | 72
  Week 15 | 73 | 55 | 70
  Week 16 | 71 | 59 | 70
  Week 17 | 69 | 59 | 67
  Week 18 | 66 | 52 | 66
  Week 19 | 64 | 54 | 67
  Week 20 | 60 | 54 | 62
  Week 21 | 56 | 54 | 61
  Week 22 | 56 | 52 | 57
  Week 23 | 51 | 54 | 63
  Week 24 | 47 | 49 | 56

13. Other Pre Specified Outcome: Time to Onset of Pain Relief
Description: Time to onset of pain relief is defined as the time from administration of study drug to the first daily pain assessment showing >30% improvement from the weekly mean of the ADP scores at baseline
Time Frame: Baseline to >30% improvement (measured up to 30 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
days | 4 [4 to 5] | 11 [7 to 24] | 3 [3 to 5]

14. Other Pre Specified Outcome: Average Weekly and Total Consumption of Rescue Medications at Each Week (Weeks 1-24)
Time Frame: Weeks 1-24
Measure: Least Squares Mean (Standard Error); unit: tablets (1 tablet = 500 mg)
Arm/Group | FX006 32 mg | Placebo | TCA IR 40 mg
Number analyzed (Participants) | 161 | 162 | 161
tablets (1 tablet = 500 mg)
  Week1 | 1.01 (0.140) | 1.31 (0.139) | 1.10 (0.140)
  Week 2 | 0.69 (0.140) | 1.39 (0.139) | 1.00 (0.140)
  Week 3 | 0.69 (0.140) | 1.35 (0.139) | 1.02 (0.140)
  Week 4 | 0.58 (0.140) | 1.28 (0.139) | 0.90 (0.140)
  Week 5 | 0.60 (0.140) | 1.21 (0.139) | 0.83 (0.140)
  Week 6 | 0.56 (0.140) | 1.24 (0.140) | 0.87 (0.140)
  Week 7 | 0.60 (0.141) | 1.19 (0.140) | 0.89 (0.140)
  Week 8 | 0.63 (0.141) | 1.24 (0.140) | 0.85 (0.140)
  Week 9 | 0.66 (0.141) | 1.11 (0.140) | 0.91 (0.140)
  Week 10 | 0.67 (0.141) | 1.21 (0.140) | 1.01 (0.140)
  Week 11 | 0.73 (0.141) | 1.12 (0.140) | 0.89 (0.140)
  Week 12 | 0.62 (0.141) | 1.13 (0.141) | 0.93 (0.140)
  Week 13 | 0.68 (0.141) | 1.14 (0.141) | 0.97 (0.140)
  Week 14 | 0.67 (0.142) | 1.18 (0.141) | 0.98 (0.141)
  Week 15 | 0.67 (0.142) | 1.25 (0.141) | 0.90 (0.141)
  Week 16 | 0.71 (0.142) | 1.15 (0.141) | 0.93 (0.141)
  Week 17 | 0.82 (0.142) | 1.17 (0.141) | 0.95 (0.141)
  Week 18 | 0.87 (0.143) | 1.15 (0.142) | 1.08 (0.141)
  Week 19 | 0.71 (0.142) | 1.23 (0.141) | 0.98 (0.141)
  Week 20 | 0.69 (0.142) | 1.22 (0.141) | 0.94 (0.141)
  Week 21 | 0.92 (0.143) | 1.23 (0.142) | 1.02 (0.141)
  Week 22 | 0.98 (0.143) | 1.21 (0.142) | 0.98 (0.141)
  Week 23 | 0.94 (0.143) | 1.20 (0.142) | 0.97 (0.141)
  Week 24 | 0.95 (0.144) | 1.18 (0.142) | 1.04 (0.141)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline Day 1 (following IA administration) through 24 weeks
Arm/Group | FX006 32mg | Placebo | TCA IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/162 | 0/161
Serious Adverse Events (participants affected / at risk) | 5/161 | 3/162 | 4/161
Other Adverse Events (participants affected / at risk) | 51/161 | 49/162 | 50/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32mg (N=161) | Placebo (N=162) | TCA IR 40 mg (N=161)
Pneumonia: (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia: (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Seizure Tonic Clonic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Unstable Angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32mg (N=161) | Placebo (N=162) | TCA IR 40 mg (N=161)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 20 (20) | 12 (12)
Headache (Vascular disorders) | 14 (14) | 13 (13) | 15 (15)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9) | 12 (12)
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (7) | 11 (11)

LIMITATIONS AND CAVEATS:
Subsequent to completion of clinical studies extensive testing was performed to assess the actual FX006 dose delivered. It was determined that the FX006 delivered dose to the patient from an FX006 40 mg vial is 32 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other